CLINICAL TRIAL: NCT00560196
Title: Pain, Anxiety and Depression in Patients With Panic Anxiety Disorders Without Pain or Depression Without Pain Compared With Healthy Volunteers
Brief Title: Pain Processing in Anxiety and Depression
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: PAD2007LG
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2009-08

CONDITIONS: Pain; Anxiety; Depression
Keywords: Neuropathic pain; Chronic pain; Depression; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression; Neuralgia; Chronic Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Patients with panic anxiety disorder without pain
  Interventions: Other: Observation
- 2: Patients with depression without pain
  Interventions: Other: Observation
- 3: Healthy controls
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
The purpose of the study is to investigate pain, anxiety and depression in patients with panic anxiety disorders without pain or depression without pain compared with healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Patients with panic disorder or depression

Exclusion Criteria:

* Treatment with antidepressants, anticonvulsants or any other pain medication except paracetamol, SSRI and benzodiazepines
* Serious or unstable medical disease
* Prior or present diagnosis of mania, bipolar or psychotic disorder, delirium, suicidal, drug and alcohol dependence, severe agitation
* Patients who cannot cooperate and do not understand Danish

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic Primary care clinic Community sample
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Quantitative sensory testing | 3-4 hours

SECONDARY OUTCOMES:
Symptom checklist 92 | 3-4 hours
Hamilton Depression and Anxiety Rating Scale | 3-4 hours
Major Depression Inventory | 3-4 hours
GAD-10 Anxiety Scale | 3-4 hours
Health Survey SF-36 | 3-4 hours
McGill Pain Questionnaire | 3-4 hours
Sweat test | 3-4 hours
Heart rate variability testing | 3-4 hours
Coping Strategy Questionnaire | 3-4 hours
Pain Catastrophizing Scale | 3-4 hours
Pain rating (VAS) | 3-4 hours
Interview | 3-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lise Gormsen, MD, Principal Investigator — Danish Pain Research Center, Aarhus University Hospital
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark